CLINICAL TRIAL: NCT03546374
Title: Irrigated Radio Frequency Ablation to Terminate Non-Paroxysmal Atrial Fibrillation (Terminate AF Study)
Brief Title: Medtronic Terminate AF Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Surgery (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT17066ECT001
Record Dates: First submitted 2018-05-09; First posted 2018-06-06 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Persistent Atrial Fibrillation; Longstanding Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Primary Cohort (Experimental): Patients with a history of persistent atrial fibrillation and long-standing persistent atrial fibrillation (non-paroxysmal atrial fibrillation) who are undergoing concomitant cardiac surgery
  Interventions: Procedure: Surgical Ablation; Device: Cardioblate and Cryoflex hand held devices

INTERVENTIONS:
Procedure: Surgical Ablation — In addition to the concomitant surgery, subjects are required to have amputation or closure (with sutures or ligation) of the left atrial appendage.The Cox Maze IV lesion set is required to be performed.
Device: Cardioblate and Cryoflex hand held devices — The Cardioblate hand held devices consist of the Cardioblate iRF and Cryo surgical ablation devices.

SUMMARY:
The purpose of this study is to demonstrate the safety and effectiveness of the Cardioblate iRF and CryoFlex hand held devices for the treatment of non-paroxysmal atrial fibrillation (AF).

DETAILED DESCRIPTION:
This is a multi-center, single-arm, prospective, non-randomized, interventional study. A maximum of 160 subjects will be treated at up to 25 centers in the United States (US). The study will include male and female patients with a history of non-paroxysmal atrial fibrillation who are undergoing concomitant cardiac surgery. Subjects will be followed and assessed after procedure and for 12 months.

The purpose of this study is to evaluate the safety and effectiveness of the Cardioblate Surgical Ablation iRF and CryoFlex hand held devices to support an indication expansion to include treatment of persistent atrial fibrillation and long-standing persistent atrial fibrillation (non-paroxysmal atrial fibrillation) to the product labeling.

ELIGIBILITY:
Inclusion Criteria:

* History of non-paroxysmal AF (persistent or longstanding persistent)
* Concomitant indication for non-emergent open-heart surgery, eg,

  1. Coronary artery bypass grafting
  2. Valve repair or replacement
* Able to take the anticoagulant warfarin or novel oral anticoagulants (NOAC)

Exclusion Criteria:

* Wolff-Parkinson-White syndrome
* New York Heart Association (NYHA) Class = IV
* Left Ventricular Ejection Fraction ≤ 30%
* Need for emergent cardiac surgery (ie, cardiogenic shock) or redo open heart surgery
* Previous AF ablation, atrioventricular (AV) -nodal ablation, or surgical Maze procedure
* Contraindication for anticoagulation therapy
* Left atrial diameter > 6.0 cm
* Preoperative need for an intra-aortic balloon pump or intravenous inotropes
* Renal failure requiring dialysis or hepatic failure
* Life expectancy of less than 1 year
* Predicted risk of operative mortality >10% as assessed by STS Risk Calculator
* Pregnancy or desire to be pregnant within 12 months of the study treatment
* Current diagnosis of active systemic infection
* Active endocarditis
* Documented MI 30 days prior to study enrollment
* Current or planned participation in an investigational or observational drug or device trial related to the treatment of atrial arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Composite acute major adverse event rate | 30-days post-procedure or hospital discharge (whichever is longer)
  Composite acute major adverse event rate including: Atrial tears, Esophageal injury, Excessive bleeding, Mediastinitis, Myocardial infarction (MI), Pulmonary embolism, Peripheral arterial embolism, Stroke, Transient ischemic attacks (TIA), Death.
Freedom from Atrial Fibrillation (AF)/Atrial Flutter (AFL)/Atrial Tachycardia (AT) | 6-months post-procedure to 12-months post-procedure
  Freedom from AF/AFL/AT of 30 seconds or greater duration on Holter, and 10 seconds on 12-lead ECG after removal from antiarrhythmic drug (AAD) therapy.

SECONDARY OUTCOMES:
Composite acute major adverse event rate (Safety) | 6-months post-procedure
  Composite acute major adverse event rate at 6 months post-procedure (as defined above)
Composite acute major adverse event rate (Safety) | 12-months post-procedure
  Composite acute major adverse event rate at 12 months post-procedure (as defined above)
Percentage of new permanent pacemaker implantation (Safety) | 12-months post-procedure
  Percentage of new permanent pacemaker implantation presented by indication
Acute procedural success (Efficacy) | During index procedure
  Acute procedural success (pulmonary vein isolation)
Freedom from AF/AFL/AT after removal of AAD therapy through 6-months post-procedure (Efficacy) | 6-months post-procedure
  Freedom from AF/AFL/AT of 30 seconds or greater duration after removal from AAD therapy as assessed from the end of the 3-month blanking period through 6 months post-procedure
Freedom from AF/AFL/AT through 6-months post-procedure (Efficacy) | 6-months post-procedure
  Freedom from AF/AFL/AT of 30 seconds or greater duration regardless of AAD status through 6 months post-procedure
Freedom from AF/AFL/AT through 12-months post-procedure (Efficacy) | 12-months post-procedure
  Freedom from AF/AFL/AT of 30 seconds or greater duration regardless of AAD status through 12 months post-procedure
Atrial Fibrillation Effect on QualiTy-of-life (AFEQT) Quality of Life Score over time (Efficacy) | 12-months post-procedure
  Characterization of quality of life scores over time as assessed by AFEQT questionnaire.
  AFEQT overall score ranges from 0-100. Zero corresponds to complete disability and 100 corresponds to no disability.
  The means, medians, standard deviations, interquartile ranges, minima, and maxima will be provided for the quality of life scores by visit interval.
SF-12 Health Survey (SF-12) Quality of Life Score over time (Efficacy) | 12-months post-procedure
  Characterization of quality of life scores over time as assessed by SF-12 questionnaire.
  SF-12 overall score ranges from 0-100. Zero indicates the lowest level of health measured by the scale and 100 indicates the highest level of health.
  The means, medians, standard deviations, interquartile ranges, minima, and maxima will be provided for the quality of life scores by visit interval.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph J Damiano, MD, Principal Investigator — Washington University School of Medicine
Locations (15):
- United States (15):
  - Stanford Hospitals and Clinic, Palo Alto, California
  - Adventist Health St. Helena, St. Helena, California
  - Hartford Healthcare, Hartford, Connecticut
  - St Vincent Heart Center of Indiana, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Corewell Health, Grand Rapids, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - ProMedica Toledo, Toledo, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Intermountain Medical Center, Murray, Utah
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Virginia Mason Heart Institute, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - St. Joseph Medical Center, Tacoma, Washington